CLINICAL TRIAL: NCT03749395
Title: Ultrasound Guided Erector Spinae Block for Postoperative Analgesia in Thoracotomy Patients : A Prospective, Randomized, Observer-Blind,Controlled Clinical Trial
Brief Title: Ultrasound Guided Erector Spinae Block for Postoperative Analgesia in Thoracotomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, mohammed gomaa sobhy, Ultrasound Guided Erector Spinae Block for Postoperative Analgesia in Thoracotomy patients : A Prospective, Randomized, Observer-Blind,Controlled Clinical Trial, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Erector spinae block
Record Dates: First submitted 2018-11-13; First posted 2018-11-21 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two parallel arms. One group will receive erector spinae plane block, and the other will receive nothing.
Who Masked: Outcomes Assessor
Masking Description: The practitioner and the patient are not blinded.The outcomes assessor will not know which group each patient is in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block group (Active Comparator): * The Erector Spinae Plane block will be done as follow,the patient will be placed in a sitting position and the ultrasound probe will be placed in a longitudinal orientation 3 cm lateral to the T5 spinous process. Three muscles were identified superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae . the needle will be inserted in a cephalad-to-caudad direction until the tip lay deep to erector spinae muscles, as evidenced by visible linear spread of fluid beneath muscle upon injection . A total of 20 mL of 0.25% bupivacaine will be injected here.
  * All patients will receive general anesthesia as described in conventional group
  Interventions: Procedure: Erector Spinae Plane Block
- Conventional group (No Intervention): * Nothing will be injected
  * All patients will receive pre-oxygenation with O2 100% for 3 min. Anesthesia will be induced by using fentanyl 1μg/kg, propofol 1.5-2 mg/kg and atracurium 0.5 mg/kg will be used for muscle relaxation. Anesthesia will be maintained by controlled ventilation with oxygen and air (50:50) with target of EtCo2≈ 35-40 mmHg, isoflurane 1:1.5 minimum alveolar concentration (MAC), 0.5μg/kg fentanyl will be given intraoperative when either heart rate or Non Invasive Blood Pressure report an increase by more than 20% of the basal records. Anesthesia will be discontinued and tracheal extubation will be done once patient fulfilled the extubation criteria.

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — The patient will be placed in a sitting position and the ultrasound probe will be placed in a longitudinal orientation 3 cm lateral to the T5 spinous process. Three muscles were identified superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae . the needle will be inserted in a cephalad-to-caudad direction until the tip lay deep to erector spinae muscles, as evidenced by visible linear spread of fluid beneath muscle upon injection . A total of 20 mL of 0.25% bupivacaine will be injected here.
  Arms: Erector Spinae Plane Block group

SUMMARY:
aim of this study is to assess and compare between the efficacy of the new U/S guided erector spinae plane block (ESP) and the conventional methods of systemic analgesics in adult patients scheduled for elective thoracotomy surgery.

DETAILED DESCRIPTION:
Thoracotomy is considered the most painful of surgical procedures and providing effective analgesia is the onus for all anesthetists. Ineffective pain relief impedes deep breathing, coughing, and remobilization culminating in atelectasis and pneumonia.The erector spinae plane (ESP) block is a newly-described technique for treating thoracic pain, and has several advantages that make it an attractive alternative to these more invasive procedures.Ultrasound guided erector spinae (ESP) block is a regional anesthesia technique, recently described by (Forero; et al.) for use in thoracic neuropathic pain. ESP block is reported to lead to analgesic effect on somatic and visceral pain by effecting the ventral rami and rami communicantes that include sympathetic nerve fibers, as LA spreads through the paravertebral space . When performed bilaterally it has been reported to be as effective as thoracic epidural analgesia.ESP block leads to effective postoperative analgesia when performed at T 4-5 level for breast and thoracic surgery. The ESP block , will be performed as follow:The patient will be placed in a sitting position and the ultrasound probe will be placed in a longitudinal orientation 3 cm lateral to the T5 spinous process. Three muscles were identified superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae . the needle will be inserted in a cephalad-to-caudad direction until the tip lay deep to erector spinae muscles, as evidenced by visible linear spread of fluid beneath muscle upon injection . A total of 20 mL of 0.25% bupivacaine will be injected here.

ELIGIBILITY:
Inclusion Criteria:

* patients aged >18 years
* American Society of Anesthesiologists Physical Status I or IV scheduled for elective thoracotomy

Exclusion Criteria:

* Refusal of the patient to provide written consent
* history of relevant drug allergy
* age less than 18
* obesity BMI > 40 kg/m2
* infection of the skin at the site of needle puncture area
* coagulopathy
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
24 hours morphine consumption | 24 hours postoperative
  total morphine consumption in both groups will be assessed in the postoperative period

SECONDARY OUTCOMES:
The quality of analgesia based on visual analogue scale (VAS) pain scores. | every 6 hours for 24 hours
  VAS score will be obtained in the postoperative period at preset time intervals.Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.No pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Side effects of opioid usage | 2, 6, 12, 24 hours postoperative
  Any evidence of opioid-related morbidity or adverse effects eg. nausea,vomiting,pruritus.These effects will be assessed by questionnaire.
Procedural morbidity | 2, 6, 12, 24 hours postoperative
  Any evidence of procedure-related morbidity

CONTACTS AND LOCATIONS:
Overall Officials: faculty of medicine, Study Director — faculty of medicine
Locations (1):
- Banha University Hospital, Banhā, Egypt

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016